CLINICAL TRIAL: NCT06956911
Title: Effect of Early Low Resisted Exercise With Blood Flow Restriction on Pulmonary Function in Post Cardiac Surgery Patient
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Toaa Mamdouh Makram, physical therapist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC\012\005679
Record Dates: First submitted 2025-04-16; First posted 2025-05-04 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Coronary Artery Bypass Grafting; Post Coronary Artery Bypass Grafting
Keywords: Post Coronary Artery Bypass Grafting

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- study group (Experimental): Traditional cardiac rehabilitation with early low resisted exercise with blood flow restriction
  Interventions: Device: traditional cardiac rehabilitation with early low resisted exercise with blood flow restriction
- control group (Active Comparator): Traditional cardiac rehabilitation only
  Interventions: Device: traditional cardiac rehabilitation

INTERVENTIONS:
Device: traditional cardiac rehabilitation with early low resisted exercise with blood flow restriction — Traditional cardiac rehabilitation and early low resisted exercise with 0.5 kilogram in form of bilateral upper limb exercise (elbow flexion and extension,wrist flexion and extension ) with external pressure applied with pressure cuff which determined by 40% of systolic blood pressure which applied on the proximal part of the arm,the frequency of exercise is once per day for 14 consecutive day and intensity determined by rate of perceived exertion scale
  Arms: study group
Device: traditional cardiac rehabilitation — Diaphragmatic and costal breathing exercise, active assisted to active range of motion,percussion,splinted cough,early mobility, upper limb exercise with breathing and incentive spirometer
  Arms: control group

SUMMARY:
After cardiac surgery Patients present a loss of exercise capacity, muscle mass, and quality of life Cardiopulmonary rehabilitation aims to reduce the loss of muscle strength, size and increase cardiopulmonary function so that quality of life is maintained as much as possible after open-heart surgeries. Traditionally, cardiac rehabilitation consist of low-intensity aerobic exercise. Therefore, cardiac rehabilitation should include not only aerobic but also resistance training (RT),. A safe and effective version of RT is needed that can still improve muscle strength and size in patients early after cardiac surgery,It is found that BFR can achieve the same result with low intensity which is suitable for patient post cardiac surgery,so the result of this study will provide a safe resisted exercise useful for post cardiac surgery patient

ELIGIBILITY:
Inclusion Criteria:

* Male patient aged from 45-60
* Elective open heart surgery via median sternotomy
* Post operative, extubated post open heart surgery, who can follow the instructions and sign the consent form
* Hemodynamic stability
* Neurological stability

Exclusion Criteria:

* Still on mechanical ventilation more than 48 hours
* Neuromuscular diseases
* Rheumatoid arthritis
* Coagulopathy
* Chronic Obstructive Pulmonary Disease (COPD)
* Cardiac arrhythmias

Ages: 45 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-11-07 (Actual); Primary Completion 2025-03-20 (Actual); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
pulmonary function test, parameters that be measured is FVC and will be expressed as % of the predicted value for age,height,weight and sex and FEV1 and will be expressed as % of the predicted value of age ,sex,weight and height | fourteen days
  parameters that be measured is FVC and will be expressed as % of the predicted value for age, height ,weight and sex and FEV1 and will be expressed as % of the predicted value of age ,sex, weight and height
Hand grip strength | fourteen days
  measure hand grip strength by hand held dynamometer (digital apperatus) expressed by kilogram
c-reactive protein lab | fourteen days
Functional capacity | fourteen days ,first measure will be at the session of assessment and last measure will be at the end of treatment program after fourteen days
  measure functional capacity by six minute walk test by calculate the total distance covered by the patient expressed by meters

CONTACTS AND LOCATIONS:
Locations (1):
- National heart institute, Cairo, Cairo Governorate, Egypt